CLINICAL TRIAL: NCT04533399
Title: A Phase 2A/B, Randomized, Observer-blinded, Placebo-controlled Study to Evaluate the Efficacy, Immunogenicity, and Safety of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine (SARS-CoV-2 rS) With Matrix-M1™ Adjuvant in South African Adult Subjects Living Without HIV; and Safety and Immunogenicity in Adults Living With HIV
Brief Title: A Study Looking at the Effectiveness and Safety of a COVID-19 Vaccine in South African Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-501
Record Dates: First submitted 2020-08-28; First posted 2020-08-31 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (HIV negative) 5 μg SARS-CoV-2 rS/Matrix-M1 Adjuvant (Experimental): 2 doses of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M1 adjuvant (co-formulated), 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant
- Cohort 1 (HIV negative) Placebo (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21.
  Interventions: Other: Placebo
- Cohort 2 (HIV positive) 5 μg SARS-CoV-2 rS/Matrix-M1 Adjuvant (Experimental): 2 doses of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M1 adjuvant (co-formulated), 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant
- Cohort 2 (HIV positive) Placebo (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Days 0 and 21.
  Other Names: NVX-CoV2373
  Arms: Cohort 1 (HIV negative) 5 μg SARS-CoV-2 rS/Matrix-M1 Adjuvant; Cohort 2 (HIV positive) 5 μg SARS-CoV-2 rS/Matrix-M1 Adjuvant
Other: Placebo — Alternating intramuscular (deltoid) injections of placebo (0.5 mL) on Days 0 and 21.
  Other Names: Sodium chloride 0.9% (BP, sterile)
  Arms: Cohort 1 (HIV negative) Placebo; Cohort 2 (HIV positive) Placebo

SUMMARY:
This is a study to evaluate the effectiveness and safety of a coronavirus disease 2019 (COVID-19) vaccine called SARS-CoV-2 rS with Matrix-M1 adjuvant in a minimum of approximately 2,960 to a maximum of approximately 4,164 healthy HIV-negative (HIV-) adult participants and in approximately 240 medically stable HIV-positive (HIV+) adult participants in up to 15 sites across South Africa. A vaccine causes the body to have an immune response that may help prevent the infection or reduce the severity of symptoms. An adjuvant is something that can make a vaccine work better. This study will look at the protective effect, body's immune response, and safety of SARS-CoV-2 rS with Matrix-M1 adjuvant in these study populations. Participants in the study will randomly be assigned to receive SARS-CoV-2 rS with Matrix-M1 adjuvant or placebo. Each participant in the study will receive a total of 2 intramuscular injections over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Adult male and female aged ≥ 18 to < 65 years at screening for Cohorts 1 and 2 and Adult male or female aged ≥ 65 to < 85 years at screening for Cohort 1 only.
* Body mass index (BMI) of 17 to 40 kg/m².
* Provides informed consent prior to study participation and is willing to comply with study procedures, including potential home visits.
* Women of child-bearing potential must agree not to have sexual intercourse with men, or must consistently use an agreed method of contraception from at least 21 days prior to enrolment in the study, through 6 months after the last vaccination.

HIV-negative subjects only:

* Documentation of HIV-negative test result by a method approved in South Africa.
* Healthy at study screening, as determined by the investigator.

HIV-positive subjects only:

* Documentation of HIV-positive test result by a method approved in South Africa.
* Receiving highly active antiretroviral therapy (HAART) and has been using the same regimen for at least 8 weeks before screening. Changes in antiretroviral dosage within 8 weeks of entering the study are allowed, as are exchanges in pharmacological formulations.
* Medically stable at screening, as determined by the investigator, and free of opportunistic infections in the 1 year prior to first study vaccination.
* Have a HIV-1 viral load < 1000 copies/mL within 45 days of randomization in the study.

Exclusion Criteria:

* Any current acute illness requiring medical or surgical care, or chronic illness (excluding HIV in HIV-positive subjects) that requires changes in medication in the past 2 months indicating that chronic illness/disease is not stable.
* Chronic disease, including:

  1. Hypertension (elevated blood pressure [BP]) ≥ grade 2 (systolic BP ≥ 160 mmHg; and/or diastolic BP ≥ 100 mmHg) according to the South African Hypertension Society's Practice Guidelines. NOTE: Hypertension [elevated BP] ≤ grade 1 (systolic BP ≤ 159 mmHg; diastolic BP ≤ 99 mmHg) according to the South African Hypertension Society's Practice Guidelines is NOT exclusionary;
  2. Congestive heart failure with a history of an acute exacerbation of any severity in the prior 2 years;
  3. Chronic obstructive pulmonary disease (COPD) with a history of an acute exacerbation of any severity in the past 2 years;
  4. Evidence of unstable coronary artery disease in the past 3 months, as determined by the investigator; NOTE: Stable coronary heart disease is NOT exclusionary.
  5. Asthma requiring regular/chronic control medication (eg, short-acting beta2-agonist [SABA] > 2 days per week; or any chronic use of inhaled corticosteroids [ICS], long-acting beta2-agonist [LABA], leukotriene receptor antagonist [LTRA], or oral corticosteroids), and/or worsening of asthma symptoms in the past 3 months; NOTE: Asthma not requiring regular/chronic control medication, and not requiring SABA > 2 days per week, and not demonstrating worsening of symptoms in the past 3 months, will NOT be excluded.
  6. Type 1 or 2 diabetes (adult onset) requiring treatment with insulin; NOTE: Non-insulin dependent type 2 diabetes is NOT exclusionary.
  7. Chronic kidney disease/renal insufficiency;
  8. Chronic gastrointestinal and hepatic diseases;
  9. Chronic neurological diseases (such as multiple sclerosis, dementia, transient ischemic attacks, Parkinson's disease, degenerative neurological conditions, neuropathy, or epilepsy), or a history of stroke within 12 months with residual symptoms, or previous neurological disorder within 12 months with residual symptoms; NOTE: History of migraine or chronic headaches, or nerve root compression that have been stable on treatment for the last 4 weeks are NOT exclusionary.
* Participation in research involving an investigational product (drug/biologic/device) within 45 days prior to first study vaccination.
* Prior receipt of investigational or approved COVID-19 vaccine at any time.
* History of a diagnosis of suspected or confirmed COVID-19.
* Received influenza (flu) vaccination within 14 days prior to first study vaccination; or any other vaccine within 4 weeks prior to first study vaccination; or planned vaccination with 5 weeks after first study vaccination.
* Any autoimmune or immunodeficiency disease/condition (excluding HIV in HIV-positive patients).
* Chronic (more than 14 days continuous) administration of immunosuppressant, systemic glucocorticosteroids, or other immune-modifying drugs within 90 days prior to first study vaccination (excluding HAART in HIV-positive subjects). NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination (excluding HAART in HIV-positive subjects).
* Acute respiratory and/or non-respiratory illness consistent with potential COVID-19, concurrent with or within 14 days prior to first study vaccination, or documented temperature of > 38°C during this period.
* Known blood clotting disorder.
* Active cancer (malignancy) within 3 years prior to first study vaccination (with the exception of adequately treated non-melanoma skin cancers, as assessed by the investigator).
* Any known allergies to products contained in the investigational product, or latex allergy, or any history of anaphylaxis in relation to any previous vaccination.
* Women who are breastfeeding or who are pregnant at the time of screening, or plan to become pregnant within the first 6 months of the study.
* History of alcohol abuse or drug addiction within 2 years prior to the first study vaccination.
* Any condition (other than HIV in HIV-positive subjects) that, in the opinion of the investigator, would pose a health risk to the subject if they participate in the study, or could interfere with evaluation of the study vaccine or interpretation of study results.
* Study team member or first-degree relative of any study member.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4422 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Cohort 1: HIV- Participants with Symptomatic Mild, Moderate, or Severe COVID-19 | Day 28 to Day 386
  Number of human immunodeficiency virus negative (HIV-) participants with first occurrence of positive (+) polymerase chain reaction (PCR), (+) PCR-confirmed, SARS-CoV-2 illness with symptomatic mild, moderate, or severe COVID-19 assessed from Day 28 (7 days after second vaccination dose) through the length of the study.
Cohort 2: HIV + Participants with Symptomatic Mild, Moderate, or Severe COVID-19 | Day 28 to Day 386
  Number of HIV+ participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with symptomatic mild,moderate or severe COVID-19 assessed from Day 28 (7 days after second vaccination) through the length of the study.
Cohort 1: HIV- Participants with Solicited Adverse Events (AEs) | 28 days
  Number of HIV- participants with solicited AEs, local and systemic, for 7 days following each vaccination (Days 0 and 21) by severity score, duration, and peak intensity.
Cohort 1: HIV- Participants with Unsolicited AEs | 35 days
  Number of HIV- participants with unsolicited AEs (eg, treatment-emergent, serious, suspected unexpected serious, those of special interest, MAAEs) through Day 35 by Medical Dictionary for Regulatory Activities (MedDRA) classification, severity score, and relatedness.
Cohort 2: HIV+ Participants with Solicited AEs | 28 days
  Number of HIV+ participants with solicited AEs, local and systemic, for 7 days following each vaccination (Days 0 and 21) by severity score, duration, and peak intensity.
Cohort 2: HIV+ Participants with Unsolicited AEs | 35 days
  Number of HIV+ participants with unsolicited AEs (eg, treatment-emergent, serious, suspected unexpected serious, those of special interest, MAAEs) through Day 35 by MedDRA classification, severity score, and relatedness.
Cohort 2: Serum Immunoglobulin G (IgG) Antibody Levels Expressed as Geometric Mean Titers (GMTs) | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMTs at Day 35.
Cohort 2: Serum IgG Antibody Levels Expressed as Geometric Mean Fold Rises (GMFRs) | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Day 35.
Cohort 2: Serum IgG Antibody Levels Expressed as Seroconversion Rates (SCRs) | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCR at Day 35. SCR is defined as the percentage of participants with a post-vaccination titer ≥ 4 fold over naïve background and ≥ 2 fold over pre existing titer.
Healthcare Worker Expansion (Cohort 3): Participants with AESI's | Day 35
  Number of healthy adult HCW, with AESIs for 14 days post second vaccination (Day 35) by severity score, duration, and peak intensity.
Healthcare Worker Expansion (Cohort 4): Participants with AESI's | Day 70
  Number of healthy adult HCW, with AESIs for 14 days post second vaccination (Day 70) by severity score, duration, and peak intensity.

SECONDARY OUTCOMES:
Cohort 1: HIV- Participants with Individual Strata of Symptomatic Virologically Confirmed, Mild, Moderate, or Severe COVID-19 | Day 28 to Day 386
  Number of HIV- participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness in terms of individual strata of symptomatic virologically confirmed, mild, moderate, or severe COVID-19.
Cohort 1: HIV- Participants with COVID-19 Requiring Hospitalization | Day 28 to Day 386
  Number of HIV- participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with COVID-19 requiring hospitalization.
Cohort 1: Incidence, Maximum Severity Score, and Symptom Duration of SARS-CoV-2 Infection by Severity Classification | Day 28 to Day 386
  Incidence, maximum severity score, and symptom duration of SARS-CoV-2 infection by classification of symptomatic virologically confirmed, mild, moderate, and/or severe disease in HIV- participants.
Cohort 1: Serum IgG Antibody Levels at Multiple Time Points Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: Serum IgG Antibody Levels at Multiple Time Points Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: Serum IgG Antibody Levels at Multiple Time Points Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV- participants. SCR is defined as the percentage of participants with a post-vaccination titer ≥ 4 fold over naïve background and ≥ 2 fold over pre-existing titer.
Cohort 1: Angiotensin-Converting Enzyme 2 (ACE2) Receptor Binding Inhibition Assay Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMTs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: ACE2 Receptor Binding Inhibition Assay Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMFRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: ACE2 Receptor Binding Inhibition Assay Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SCRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: ACE2 Receptor Binding Inhibition Assay Expressed as Seroresponse Rates (SRRs) | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SRRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants. SRR is defined as the proportion of participants with rises in titers exceeding the 95th percentile of placebo participants at the same time point and based on prior SARS-CoV-2 exposure.
Cohort 1: Neutralizing Antibody Activity Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by microneutralization assay (MN) as expressed as GMTs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: Neutralizing Antibody Activity Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as GMFRs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV-participants.
Cohort 1: Neutralizing Antibody Activity Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as SCRs (≥ 4 fold change) at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV- participants.
Cohort 1: Neutralizing Antibody Activity Expressed as SRRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as SRRs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV-participants.
Cohort 1: HIV- Participants with Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) | 386 days
  Numbers and percentages (with 95% CI) of participants with MAAEs, AESI, or SAE through End of Study by MedDRA classification, severity score, and relatedness in HIV- participants.
Cohort 2: Serum IgG Antibody Levels at Multiple Time Points Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: Serum IgG Antibody Levels at Multiple Time Points Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: Serum IgG Antibody Levels at Multiple Time Points Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs at Days 0 (baseline), 21 (post first dose), and at 3 and 6 months after the last vaccination in HIV+ participants. SCR is defined as the percentage of participants with a post-vaccination titer ≥ 4 fold over naïve background and ≥ 2 fold over pre-existing titer.
Cohort 2: ACE2 Receptor Binding Inhibition Assay Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMTs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: ACE2 Receptor Binding Inhibition Assay Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMFRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: ACE2 Receptor Binding Inhibition Assay Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SCRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: ACE2 Receptor Binding Inhibition Assay Expressed as SRRs | Day 0 to 6 months after the last vaccination
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SRRs at Days 0 (baseline), 21 (post first dose), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants. SRR is defined as the proportion of participants with rises in titers exceeding the 95th percentile of placebo participants at the same time point and based on prior SARS-CoV-2 exposure.
Cohort 2: Neutralizing Antibody Activity Expressed as GMTs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN as expressed as GMTs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: Neutralizing Antibody Activity Expressed as GMFRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as GMFRs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: Neutralizing Antibody Activity Expressed as SCRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as SCRs (≥ 4 fold change) at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: Neutralizing Antibody Activity Expressed as SRRs | Day 0 to 6 months after the last vaccination
  Neutralizing antibody activity as detected by MN expressed as SRRs at Days 0 (baseline), 35 (post second dose), and at 3 and 6 months after the last vaccination in HIV+ participants.
Cohort 2: HIV+ Participants with MAAEs, AESIs, and SAEs | 386 days
  Number of participants with MAAEs, AESI, or SAE through End of Study by MedDRA classification, severity score, and relatedness in HIV+ participants.
Cohort 2: HIV+ Participants with Symptomatic Virologically Confirmed, Mild, Moderate, or Severe COVID-19 | Day 28 to Day 385
  Counts and proportions of symptomatic virologically confirmed, mild, moderate, and severe COVID-19 outcomes in HIV+ participants as previously described in the second primary efficacy endpoint for Cohort 1 (HIV- participants).
Cohort 2: Incidence, Maximum Severity Score, and Symptom Duration of SARS-CoV-2 Infection by Severity Classification | Day 28 to Day 385
  Incidence, maximum severity score, and symptom duration of SARS-CoV-2 infection by classification of symptomatic virologically confirmed, mild, moderate, and/or severe disease in HIV+ participants.
Cohort 1: HIV- Participants with Asymptomatic, Symptomatic Mild, Moderate, or Severe COVID-19 | Day 28
  Number of HIV- participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with asymptomatic, symptomatic mild, moderate or severe COVID-19 assessed from 7 days after the second vaccine dose (eg, Day 28)
Cohort 2: HIV+ Participants with Asymptomatic, Symptomatic Mild, Moderate, or Severe COVID-19 | Day 28
  Number of HIV+ participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with asymptomatic, symptomatic mild, moderate or severe COVID-19 assessed from 7 days after the second vaccine dose (eg, Day 28)
Healthcare Worker Expansion (Cohort 3): Serum IgG Antibody Expressed as GMT | Day 35
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA using GMTs at 14 days post second vaccination (Day 35 for Cohort 3) in adult HCW.
Healthcare Worker Expansion (Cohort 3): Serum IgG Antibody Expressed as GMEU | Day 35
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as GMEU at 14 days post second vaccination (Day 35 for Cohort 3) in adult HCW.
Healthcare Worker Expansion (Cohort 3): Serum IgG Antibody Expressed as GMFR | Day 35
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as GMFR at 14 days post second vaccination (Day 35 for Cohort 3) in adult HCW.
Healthcare Worker Expansion (Cohort 3): Serum IgG Antibody Expressed as SCR | Day 35
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as SCR at 14 days post second vaccination (Day 35 for Cohort 3) in adult HCW.
Healthcare Worker Expansion (Cohort 4): Serum IgG Antibody Expressed as GMT | Day 70
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as GMT at 14 days post second vaccination (Day 70 for Cohort 4) in adult HCW.
Healthcare Worker Expansion (Cohort 4): Serum IgG Antibody Expressed as GMEU | Day 70
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as GMEU at 14 days post second vaccination (Day 70 for Cohort 4) in adult HCW.
Healthcare Worker Expansion (Cohort 4): Serum IgG Antibody Expressed as GMFR | Day 70
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as GMFR at 14 days post second vaccination (Day 70 for Cohort 4) in adult HCW.
Healthcare Worker Expansion (Cohort 4): Serum IgG Antibody Expressed as SCR | Day 70
  Serum IgG antibody levels specific for the SARS CoV 2 rS protein antigen(s) as detected by ELISA expressed as SCR at 14 days post second vaccination (Day 70 for Cohort 4) in adult HCW.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (14):
- South Africa (14):
  - ZA018, Bloemfontein, Free State of South Africa
  - ZA003, Hillbrow, Gauteng
  - Site ZA001, Johannesburg, Gauteng
  - ZA012, Johannesburg, Gauteng
  - Site ZA015, Pretoria, Gauteng
  - ZA023, Pretoria, Gauteng
  - ZA019, Durban, KwaZulu-Natal
  - ZA020, Durban, KwaZulu-Natal
  - ZA021, Durban, KwaZulu-Natal
  - ZA024, Durban, KwaZulu-Natal
  - ZA007, Thabazimbi, Limpopo
  - ZA022, Madibeng, North West
  - ZA013, Cape Town, Western Cape
  - ZA014, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhi SA, Moodley D, Hanley S, Archary M, Hoosain Z, Lalloo U, Louw C, Fairlie L, Fouche LF, Masilela MSL, Singh N, Grobbelaar C, Ahmed K, Benade G, Bhikha S, Bhorat AE, Bhorat Q, Joseph N, Dheda K, Esmail A, Foulkes S, Goga A, Oommen Jose A, Kruger G, Kalonji DJ, Lalloo N, Lombaard JJ, Lombard Koen A, Kany Luabeya A, Mngqibisa R, Petrick FG, Pitsi A, Tameris M, Thombrayil A, Vollgraaff PL, Cloney-Clark S, Zhu M, Bennett C, Albert G, Faust E, Plested JS, Fries L, Robertson A, Neal S, Cho I, Glenn GM, Shinde V; 2019nCoV-501 Study Group. Immunogenicity and safety of a SARS-CoV-2 recombinant spike protein nanoparticle vaccine in people living with and without HIV-1 infection: a randomised, controlled, phase 2A/2B trial. Lancet HIV. 2022 May;9(5):e309-e322. doi: 10.1016/S2352-3018(22)00041-8. PMID 35489376
- [Derived] Shinde V, Bhikha S, Hoosain Z, Archary M, Bhorat Q, Fairlie L, Lalloo U, Masilela MSL, Moodley D, Hanley S, Fouche L, Louw C, Tameris M, Singh N, Goga A, Dheda K, Grobbelaar C, Kruger G, Carrim-Ganey N, Baillie V, de Oliveira T, Lombard Koen A, Lombaard JJ, Mngqibisa R, Bhorat AE, Benade G, Lalloo N, Pitsi A, Vollgraaff PL, Luabeya A, Esmail A, Petrick FG, Oommen-Jose A, Foulkes S, Ahmed K, Thombrayil A, Fries L, Cloney-Clark S, Zhu M, Bennett C, Albert G, Faust E, Plested JS, Robertson A, Neal S, Cho I, Glenn GM, Dubovsky F, Madhi SA; 2019nCoV-501 Study Group. Efficacy of NVX-CoV2373 Covid-19 Vaccine against the B.1.351 Variant. N Engl J Med. 2021 May 20;384(20):1899-1909. doi: 10.1056/NEJMoa2103055. Epub 2021 May 5. PMID 33951374
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — http://www.CDC.gov/coronavirus/2019-nCoV/index.html
- See also: WHO COVID-19 treatment guidelines — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/
- See also: WHO South Africa website — https://www.afro.who.int/countries/south-africa
- See also: COVID-19 Corona Virus - Department of Health, Republic of South Africa — https://sacoronavirus.co.za/